CLINICAL TRIAL: NCT00755183
Title: A Single-Center, Double-Masked, Randomized, Vehicle Controlled Study to Evaluate the Safety and Efficacy of Testosterone 0.03% Ophthalmic Solution Compared to Vehicle for the Treatment of Meibomian Gland Dysfunction
Brief Title: Safety and Efficacy Study of a Testosterone Eye Drop for the Treatment of Meibomian Gland Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-004-16
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Meibomian Gland Dysfunction
Keywords: Meibomian Gland Dysfunction; Dry Eye Syndrome
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- testosterone ophthalmic solution (Experimental): testosterone ophthalmic solution 0.03%
  Interventions: Drug: testosterone ophthalmic solution
- vehicle (Placebo Comparator): vehicle of testosterone ophthalmic solution
  Interventions: Drug: vehicle of testosterone ophthalmic solution

INTERVENTIONS:
Drug: testosterone ophthalmic solution — testosterone ophthalmic solution for 128 days
  Arms: testosterone ophthalmic solution
Drug: vehicle of testosterone ophthalmic solution — vehicle of testosterone ophthalmic solution for 128 days
  Arms: vehicle

SUMMARY:
The objective of this study is to assess the safety and efficacy of testosterone 0.03% ophthalmic solution compared to vehicle for the treatment of meibomian gland dysfunction.

DETAILED DESCRIPTION:
Meibomian gland secretion plays a crucial role in the health of the ocular surface and function of the tear film. The lipid secreted by the meibomian glands has many crucial roles: 1) to retard evaporation from the preocular surface; 2) lower the surface tension of tears; 3) prevent spill-over of tears from the lid margin; 4) prevent the contamination of the tear film by sebaceous lipids; 5) prevent damage to the skin of the lid margin. In dry eye syndrome, blepharitis, meibomian gland dysfunction, and meibomitis the glands are the central pathophysiology of disease and thus a potential target for therapy.

ELIGIBILITY:
Inclusion Criteria (subjects must):

* Be ≥ 60 years of age
* Have a corrected visual acuity of LogMAR +0.5 (ETDRS)
* Have a documented history of Meibomian Gland Dysfunction
* Have a TFBUT ≤ 5 seconds
* Have an ocular discomfort score ≥ 1
* Have an IOP ≤ 25 mmHg at Visit 1 in both eyes
* Report use of and/or desire to use an artificial tears

Exclusion Criteria (subjects may not):

* Have contraindications to the use of the study medications
* Have a known allergy or sensitivity to the study medications
* Have any ocular infections, or active ocular inflammation
* Have used ocular medications within 24 hours prior to Visit 1
* Be a current contact lens wearer
* Require the use of any other ophthalmic medication, other than tear substitutes and study medication provided, for the duration of the trial
* Have used systemic or topical antihistamines or steroids 48 hours prior to Visit 1 or require the use of systemic or topical antihistamines or steroids during the course of the study
* Have a history of prostate cancer

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Jerome Crampton, MD, Principal Investigator — ORA, Inc.
Locations (1):
- Ophthalmic Research Associates, Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Testosterone Ophthalmic Solution: testosterone ophthalmic solution 0.03%
  Participants received 1 drop of testosterone ophthalmic solution in each eye for approximately 168 days.
- Vehicle: vehicle of testosterone ophthalmic solution
  Participants received 1 drop of vehicle of testosterone ophthalmic solution in each eye for approximately 168 days.
Period: Overall Study
Arm/Group | Testosterone Ophthalmic Solution | Vehicle
Started | 30 | 30
Completed | 23 | 24
Not Completed | 7 | 6
Not completed — Adverse Event | 5 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Administrative | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone Ophthalmic Solution | Vehicle | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 25
  >=65 years | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.57 (6.730) | 68.10 (6.764) | 68.83 (6.730)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 29 | 58
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 29 | 29 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Meibomian Gland Secretion Appearance at Visit 4 (Day 168)
Description: The average of the secretion color, quality, and viscosity of the worst gland in the worst eye. All scales were numerical analog, 0-3, where 0=normal and 3=worst.
Time Frame: 168 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone Ophthalmic Solution | Vehicle
Number analyzed (Participants) | 18 | 17
units on a scale | 0.80 (0.50) | 0.96 (0.67)

2. Primary Outcome: Ocular Discomfort Score at Visit 4
Description: Ocular Discomfort Score on a 0-4 scale where 0=none and 4=constant discomfort at Visit 4 (Day 168)
Time Frame: 168 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Testosterone Ophthalmic Solution | Vehicle
Number analyzed (Participants) | 18 | 17
score on a scale | 1.70 (0.6) | 1.33 (0.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signing of the informed consent for to the end of treatment, approximately 6 months
Arm/Group | Testosterone Ophthalmic Solution | Vehicle
Serious Adverse Events (participants affected / at risk) | 2/30 | 0/30
Other Adverse Events (participants affected / at risk) | 5/30 | 5/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Ophthalmic Solution (N=30) | Vehicle (N=30)
Essential tremor (Nervous system disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Testosterone Ophthalmic Solution (N=30) | Vehicle (N=30)
Visual acuity reduced (Eye disorders) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 3
Rhinitis (Infections and infestations) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes